CLINICAL TRIAL: NCT02157974
Title: Assessment of Hepatic Glucose and Fat Regulation in Overweight Adolescent Girls
Brief Title: Liver and Fat Regulation in Overweight Adolescent Girls
Acronym: APPLE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-0542; UL1TR001082 (NIH); K23DK107871 (NIH)
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Hepatic Steatosis; Polycystic Ovarian Syndrome; Obesity
MeSH Terms: conditions — Fatty Liver; Polycystic Ovary Syndrome; Obesity | interventions — Exenatide; penclomedine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PCOS, medication naive + Byetta (Experimental): PCOS, medication naive; 10 girls with PCOS will receive 2 doses of Byetta.
  Interventions: Drug: Byetta 5Mcg Pen Injection
- Control (No Intervention): Up to 25 girls without PCOS
- PCOS medication naive (No Intervention): Up to 45 girls with PCOS with no exposure to hormone therapy or metformin in the preceding 6 months.
- PCOS on COCPs (No Intervention): Up to 10 girls with PCOS and 6 months of therapy with combined oral contraceptives (COCPs) prior to study procedures.
- PCOS on metformin (No Intervention): Up to 10 girls with PCOS and 6 months of therapy with metformin prior to study procedures

INTERVENTIONS:
Drug: Byetta 5Mcg Pen Injection — 10 participants will receive 2 doses of Byetta, one at 7 PM the night prior to metabolic study and the second 30 min before ingestion of glucola
  Other Names: Exenatide
  Arms: PCOS, medication naive + Byetta

SUMMARY:
Women with polycystic ovarian syndrome (PCOS) have increased rates of hepatic steatosis compared to weight similar women with regular menses. It is unclear if this is related to high testosterone or insulin resistance. The investigators will assess hepatic glucose release, rates of lipolysis and hepatic de novo lipogenesis in the fasted and postprandial state to determine if alterations in the processes contribute to hepatic steatosis. Participants will be overweight, sedentary girls with or without PCOS. Those with PCOS will either be medication naive, or must be taking metformin or combined oral contraceptives (COCPs) for a period of at least 6 months prior to study procedures.

DETAILED DESCRIPTION:
Hepatic glucose release will be assessed with a stable isotope glycerol tracer, lipolysis with a glycerol tracer, and hepatic de novo lipogenesis with an acetate tracer. Data will be collected fasting and after a glucose challenge. The degree of hepatic steatosis and abdominal fat partitioning will be assessed with Magnetic Resonance Imaging (MRI), and total body composition with Dual-energy X-ray absorptiometry (DEXA).

ELIGIBILITY:
Inclusion Criteria:

* Females
* 2 years post-menarche
* BMI percentile >90%

Exclusion Criteria:

* Type 2 diabetes
* Anemia
* Liver disease
* Medications known to effect insulin sensitivity
* Cause of oligomenorrhea or hirsutism other than PCOS,
* >3 hours a week of moderate exercise.

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Cree Green, MD, PhD, Principal Investigator — Department of Endocrinology
Locations (1):
- University of Colorado Anshutz Medical Campus/Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be shared with IRB approved personnel.

REFERENCES:
- [Derived] Carreau AM, Pyle L, Garcia-Reyes Y, Rahat H, Vigers T, Jensen T, Scherzinger A, Nadeau KJ, Cree-Green M. Clinical prediction score of nonalcoholic fatty liver disease in adolescent girls with polycystic ovary syndrome (PCOS-HS index). Clin Endocrinol (Oxf). 2019 Oct;91(4):544-552. doi: 10.1111/cen.14062. Epub 2019 Aug 16. PMID 31301251
- [Derived] Simon SL, McWhirter L, Diniz Behn C, Bubar KM, Kaar JL, Pyle L, Rahat H, Garcia-Reyes Y, Carreau AM, Wright KP, Nadeau KJ, Cree-Green M. Morning Circadian Misalignment Is Associated With Insulin Resistance in Girls With Obesity and Polycystic Ovarian Syndrome. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3525-3534. doi: 10.1210/jc.2018-02385. PMID 30888398

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Up to 25 girls without PCOS.
  No participants received an intervention in this specific study.
- PCOS Medication Naive: Up to 45 girls with PCOS with no exposure to hormone therapy or metformin in the preceding 6 months.
  No participants received an intervention in this specific study.
- PCOS, Medication Naive + Byetta: PCOS, medication naive;
  These 10 participants received 2 doses of Byetta during their metabolic visit prior to the oral glucose tolerance testing.
  These participants recieved Byetta 5Mcg Pen Injection: 10 participants will receive 2 doses of Byetta, one at 7 PM the night prior to metabolic study and the second 30 min before ingestion of glucola
- PCOS on COCPs: Up to 10 girls with PCOS and 6 months of therapy with combined oral contraceptives (COCPs) prior to study procedures.
  No participants received an intervention in this specific study.
- PCOS on Metformin: Up to 10 girls with PCOS and 6 months of therapy with metformin prior to study procedures
  No participants received an intervention in this specific study.
Period: Overall Study
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin
Started | 24 | 42 | 10 | 10 | 6
Completed | 24 | 39 | 10 | 10 | 6
Not Completed | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Screen Failure | 0 | 1 | 0 | 0 | 0
Not completed — Nurse not able to place IV so unable to complete visit | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin | Total
Number analyzed (Participants) | 24 | 42 | 10 | 10 | 6 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 34 | 7 | 9 | 6 | 79
  Between 18 and 65 years | 1 | 8 | 3 | 1 | 0 | 13
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.62) | 15.9 (1.81) | 15.3 (2.16) | 15.7 (1.34) | 15.6 (1.7) | 15.62 (1.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 42 | 10 | 10 | 6 | 92
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 20 | 3 | 6 | 4 | 48
  Not Hispanic or Latino | 9 | 22 | 7 | 4 | 2 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 42 | 10 | 10 | 6 | 92

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Glucose Release
Description: Hepatic glucose release will be measured by the rate of appearance of a glucose tracer. Glucose rate of appearance reflects the amount of glucose being release by primarily the liver during fasting. A higher glucose rate of appearance is often seen with dysglycemia
Time Frame: Measured up to 4 months from enrollment
Population: Not all participants had complete data to analyze the glucose RA.
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin
Number analyzed (Participants) | 16 | 30 | 9 | 8 | 4
mg/kg/min | 1.85 (1.24) | 1.46 (0.21) | 1.54 (0.38) | 1.88 (0.49) | 1.57 (0.07)

2. Secondary Outcome: Hepatic Phosphate Concentrations
Description: Hepatic phosphate relative concentrations will be measured with 31 phosphorus magnetic resonance spectroscopy. The ratio of the following will be reported over total phosphate concentration: Phosphodiesterase (PDE), phosphomonoester (PME), Adenosine triphosphate (ATP), Inorganic Phosphate (Pi),Nicotinamide adenine dinucleotide phosphate (NADPH), Uridine diphosphate glucose (UDPG)
Time Frame: Measured up to 4 months from enrollment
Population: The phosphorus coil for the liver was purchased towards the end of the study, so not all participants had the 31p measured.
Measure: Mean (Standard Deviation); unit: ratio over total phosphate
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin
Number analyzed (Participants) | 5 | 0 | 8 | 9 | 6
ratio over total phosphate
  PDE/TP | 0.167684728 (0.056413082) |  | 0.198640255 (0.040933351) | 0.198787476 (0.045832565) | 0.186923469 (0.039481266)
  PME/TP | 0.067905319 (0.033816456) |  | 0.077949656 (0.02943916) | 0.075872089 (0.024970918) | 0.066789803 (0.036986035)
  ATP/TP | 0.592517535 (0.038294886) |  | 0.566952309 (0.061717281) | 0.565157308 (0.042119495) | 0.557277652 (0.034367129)
  Pi/TP | 0.041945761 (0.02076513) |  | 0.054581135 (0.019288097) | 0.046604505 (0.022669904) | 0.074459672 (0.021584936)
  NADPH/TP | 0.097201285 (0.043438464) |  | 0.068550332 (0.028503778) | 0.067305736 (0.033620062) | 0.074693726 (0.021031863)
  UDPG/TP | 0.032745372 (0.011777685) |  | 0.033326313 (0.014030497) | 0.046272886 (0.023894603) | 0.039855678 (0.012418624)

3. Secondary Outcome: Rates of Lipolysis
Description: Rate of lipolysis will be measured by the rate of appearance of a glycerol tracer. Glycerol rate of appearance reflects the amount of glycerol being released into the blood stream as a results of lipolysis. Higher rates of lipolysis are thought to be associated with insulin resistance.
Time Frame: Measured up to 4 months from enrollment
Population: Not all participants had complete data to analyze the glycerol RA.
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin
Number analyzed (Participants) | 18 | 32 | 10 | 10 | 6
mg/kg/min | 0.54 (0.17) | 0.49 (0.22) | 0.49 (0.24) | 0.78 (0.18) | 0.65 (0.19)

4. Secondary Outcome: Hepatic Fat Fraction
Description: Amount of fat in the liver measured by MRI and calculated via the Dixon method as the proton density hepatic fat fraction, which ranges from 0-75%. Greater than 5% is considered extra fat in the liver.
Time Frame: Measured up to 4 months from enrollment
Population: Unable to analyze 2 participants in the PCOS medication naive group. One screen failed and the second who withdrew from the study.
Measure: Mean (Standard Deviation); unit: percent fat
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin
Number analyzed (Participants) | 24 | 40 | 10 | 10 | 6
percent fat | 4.1 (3.1) | 7.6 (6.3) | 6.9 (5.3) | 6.8 (9.4) | 13.3 (12.1)

5. Secondary Outcome: Hepatic de Novo Lipogenesis
Description: Hepatic de novo lipogenesis will be measured by with an acetate tracer by mass spectroscopy. De novo lipogenesis can contribute to non-alcoholic fatty liver disease, so having a lower value is better.
Time Frame: Measured up to 4 months from enrollment
Population: Not everyone in the study received the acetate tracer. We had a problem with the analysis of the acetate tracer on 3 participants: 1 from the control group and 2 from the metformin group, so we did not obtain data for those 3 participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin
Number analyzed (Participants) | 9 | 12 | 10 | 5 | 3
mg/dL | 9.3 (5.3) | 6.6 (4.2) | 7.9 (7.2) | 18.2 (14.9) | 19.4 (17.4)

6. Other Pre Specified Outcome: Whole Body Insulin Sensitivity
Description: Participants will undergo a 75 gram oral glucose tolerance test, and whole body insulin sensitivity will be expressed as Si, calculated via the oral minimal model using SAMM II software. This software uses participant weight, glucose and insulin concentrations at various time points during the oral glucose tolerance test to calculate the participant insulin sensitivity. The higher the Si value means more insulin sensitivity.
Time Frame: Measured up to 4 months from enrollment
Population: We were unable to calculate Si for some of the participants, because we were missing some lab values that are required for the formula.
Measure: Mean (Standard Deviation); unit: dL/kg/min/μU/mL
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin
Number analyzed (Participants) | 23 | 33 | 10 | 10 | 6
dL/kg/min/μU/mL | 0.000319383 (0.00021025) | 0.00021077 (0.000275814) | 0.00033516 (0.000366279) | 0.00021791 (0.000255919) | 0.0000959833333 (0.0000414436685)

7. Other Pre Specified Outcome: Sleep Quality
Description: Apnea Hypopnea Index (AHI) will be measured using WatchPAT. In children and adolescents the scale that will be used is AHI>5 is considered mild sleep apnea. The higher the AHI, indicates more severe sleep apnea.
  The AHI is the number of times you have apnea or hypopnea during one night, divided by the hours of sleep.
  Normal sleep: An AHI of fewer than five events, on average, per hour Mild sleep apnea: An AHI of five to 14 events per hour Moderate sleep apnea: An AHI of 15 to 29 events per hour Severe sleep apnea: An AHI of 30 or more events per hour
Time Frame: Measured up to 4 months from enrollment
Population: The WatchPAT device was purchased towards the end of the study, so this was only used on a few participants for which results are reported here.
Measure: Mean (Standard Deviation); unit: Apnea Hypopnea Index
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin
Number analyzed (Participants) | 2 | 0 | 2 | 5 | 2
Apnea Hypopnea Index | 9.15 (4.71) |  | 31.25 (12.09) | 19.32 (11.85) | 19 (0.57)

8. Other Pre Specified Outcome: Sleep Duration
Description: Sleep duration will be assessed using home actigraphy using the Philips Actigraph wrist-worn watch, and collects 7 days of data.
Time Frame: Measured up to 4 months from enrollment
Population: Watch failed to record data on: 3 participants in the control group, 2 in the PCOS medication naive group, and 1 in the Byetta group. Two participants withdrew from the PCOS medication naive group.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin
Number analyzed (Participants) | 21 | 38 | 9 | 10 | 6
minutes | 430.85 (48.38) | 437.88 (49.32) | 410.3 (58) | 438.29 (49.76) | 414.87 (62.29)

ADVERSE EVENTS:
Time Frame: Measured up to 4 months from enrollment
Arm/Group | Control | PCOS Medication Naive | PCOS, Medication Naive + Byetta | PCOS on COCPs | PCOS on Metformin
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/42 | 0/10 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/42 | 0/10 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 0/24 | 0/42 | 0/10 | 0/10 | 0/6

LIMITATIONS AND CAVEATS:
Due to the Covid-19 outbreak, we were unable to enroll the last 4 participants in the PCOS on metformin arm, so the results may not reach statistical significance. We had delays in getting tracer results due to the mass spec machine being down, and once raw data was obtained, we needed to work with a mathematician to calculate the rates of appearance of the tracer results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT02157974/Prot_SAP_000.pdf